CLINICAL TRIAL: NCT05120609
Title: A Randomized, Cross-Over, Placebo-Controlled Pilot Study to Evaluate the Self-Management of Gait, Speech and Dexterity in Patients With Parkinson's Disease Using a Novel Digital Therapeutic Approach
Brief Title: Pilot Study to Evaluate the Self-Management of Gait, Speech, and Dexterity Symptoms in Parkinson's Disease Using a Smartphone Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beats Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2021-11-04; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
Keywords: Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases; Brain Diseases; Central Nervous System Diseases
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases; Brain Diseases; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Application (Experimental): Subjects will complete at-home allied health therapy exercises delivered through a smartphone application. Subjects will use the application daily for 4 weeks, each daily session takes up to 30 minutes to complete.
  Interventions: Device: Parkinson's Application
- Digital Placebo (Placebo Comparator): Subjects will have access to a digital placebo application and continue usual care.
  Interventions: Device: Digital Placebo Application

INTERVENTIONS:
Device: Parkinson's Application — The application delivers at-home, tailored allied health exercises (physiotherapy, speech and language therapy, and occupational therapy) for the gait, speech, and manual dexterity symptoms associated with Parkinson's disease.
  Arms: Parkinson's Application
Device: Digital Placebo Application — The application is designed to provide a method of capturing outcome measures without providing access to the therapy exercises.
  Arms: Digital Placebo

SUMMARY:
The purpose of this study is to evaluate the impact of a smartphone application that delivers at-home therapy exercises on patients' self-management of gait, speech, and dexterity symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 30 years of age or older,
* History of idiopathic Parkinson's Disease (Hoehn and Yahr stage of II-IV),
* Normal joint range of motion in both legs,
* Able to walk independently for 10 feet with or without an assistive device,
* Parkinson's gait and mild to moderate speech impairment,
* No history of vestibular disease,
* No evidence of dementia (MMSE ≥24),
* Clear benefit from Levodopa,
* Agrees to Beats Medical Application Privacy Policy and Terms of Use,
* Access to an iPhone 7 or higher to use the Beats Medical applications.

Exclusion Criteria:

* Medical condition for which exercise is contraindicated,
* History or evidence of neurological deficit other than Parkinson's Disease that could interfere, such as previous stroke or muscle disease,
* History or evidence of orthopaedic or muscular problems,
* Subject is currently enrolled in a study to evaluate an investigational drug or device,
* Subject unable or unwilling to provide informed consent,
* Vulnerable populations as deemed inappropriate for the study by site Principal Investigator,
* History of falls in the past 6 months,
* Pregnancy,
* Current or previous use of the Beats Medical Parkinson's application.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Velocity (m/s) | Baseline, Week 4, Week 8, Week 12
  Gait velocity on a 10-Meter Walk Test (10MWT) conducted in-clinic.

SECONDARY OUTCOMES:
Step Length (m) | Baseline, Week 4, Week 8, Week 12
  Change in Step length on a 10-Meter Walk Test (10MWT) conducted in-clinic.
Step Frequency (steps/min) | Baseline, Week 4, Week 8, Week 12
  Change in Step frequency on a 10-Meter Walk Test (10MWT) conducted in-clinic.
MDS-UPDRS Total Score for Part II Item 2.1 + Part III Item 3.1 | Baseline, Week 4, Week 8, Week 12
  Movement Disorders Society Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is designed to monitor the burden and extent of Parkinson's disease. The MDS-UPDRS is divided into 4 parts: (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. In each part, all items are rated on a scale from 0-4, with higher scores reflecting greater severity.
  The sum of items 2.1 (Speech) and Part III 3.1 (Speech) will be used to calculate a total score to assess speech abilities.
MDS-UPDRS Total Score for Part II Item 2.7 + Part III Item 3.4 + Part III 3.5 | Baseline, Week 4, Week 8, Week 12
  The sum of items 2.7 (handwriting), 3.4 (finger tapping), and 3.5 (hand movements) will be used to calculate a total score to assess manual dexterity. All items are rated on a scale from 0-4, with higher scores reflecting greater severity.
MDS-UPDRS Part II Total Score | Baseline, Week 4, Week 8, Week 12
  For MDS-UPDRS Part II (motor experiences of daily living) scores, the scale range for Part II Total Score is 0-52, with higher scores reflecting greater severity.
Daily steps | Week 1,2,3,4,5,6,7,8
  Physical activity will be assessed by the relative change in daily steps recorded by the in-device sensors in the smartphone.

OTHER OUTCOMES:
Average duration (seconds) of sustained vowel phonation | Baseline, Week 4, Week 8, Week 12
  Change in the average duration of sustained vowel phonation on a smartphone-based speech assessment conducted in-clinic.
Time taken to complete a smartphone-based 9-Hole Peg Test (seconds) | Baseline, Week 4, Week 8, Week 12
  Change in time taken to complete a smartphone-based 9-Hole Peg Test conducted in-clinic.
Total Distance (m) walked on a smartphone-based 2-minute walk test (2MWT) | Baseline, Week 4, Week 8, Week 12
  Change in total distance walked on a smartphone-based at-home 2-minute walk test (2MWT).
Gait velocity (m/s) on a smartphone based 2-minute walk test (2MWT) | Baseline, Week 4, Week 8, Week 12
  Chance in gait velocity on a smartphone-based at-home 2-minute walk test (2MWT).
Step frequency (steps/min) on a smartphone-based 2-minute walk test (2MWT) | Baseline, Week 4, Week 8, Week 12
  Change in step frequency on a smartphone-based at-home 2-minute walk test (2MWT).

CONTACTS AND LOCATIONS:
Locations (1):
- Meridian Clinical Research, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No